CLINICAL TRIAL: NCT01832779
Title: Prospective Evaluation of the Clinical Utility of Peroral Endoscopic Myotomy (POEM)
Brief Title: Peroral Endoscopic Myotomy (POEM) for the Treatment of Achalasia
Acronym: POEM
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201300104
Record Dates: First submitted 2013-04-02; First posted 2013-04-16 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Achalasia
Keywords: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Achalasia subjects: Information about teh subject's medical history, leading up to the need for an Achalasia treatment, the procedure itself and how the subject does after the procedure, including after the subject gets home, will be collected. This will be done by gathering relevant information from the subject's medical chart and/or by talking with the subject prior to and after the subject's medical procedures. There are no specific study procedures or tests. All information collected is part of the subject's medical care and will be collected even if the subject is not in the study.
  Interventions: Other: Achalasia subjects

INTERVENTIONS:
Other: Achalasia subjects — Information about the subject's medical history, leading up to the need for an Achalasia treatment, the procedure itself and how the subject does after the procedure, including after the subject's gets home, will be collected. This will be done by gathering relevant information from the subject's medical chart and/or by talking with the subject prior to and after your medical procedures. There are no specific study procedures or tests. All information collected is part of the subject's medical care and will be collected even if the subject is not in the study.
  Other Names: Peroral Endoscopic Myotomy

SUMMARY:
Achalasia is a chronic disease of altered esophageal motility with resulting functional obstruction to the passage of food leading to poor quality of life and significant morbidity. The two main treatments available in the US are endoscopic balloon dilation and surgical myotomy. Each therapy has advantages and drawbacks and at present both are considered a first choice approach depending on patient preferences and local expertise. Surgical myotomy provides long lasting improvement in dysphagia but even when done laparoscopically is invasive and complex. Extensive acid reflux resulting in significant morbidity is routinely seen after surgical myotomy and additional anti-reflux operation is typically done at the time of the myotomy. Endoscopic balloon dilation is a simple minimally invasive outpatient procedure but improvement of symptoms tends to be shorter in duration and repeat dilations are commonly needed. Both therapies improve on dysphagia but tend to provide suboptimal control of chest pain which is one of the cardinal symptoms of achalasia.

The peroral endoscopic myotomy (POEM) was first introduced in Japan to address the suboptimal results with endoscopic balloon dilation and surgical myotomy. POEM is incisionless minimally invasive but in addition may have some further advantages over surgical myotomy including unlimited length of the myotomy with expected better control of chest pain and preservation of the anatomical anti-reflux barrier (angle of His and the cruse of the diaphragm) with expected lower incidence of acid reflux.

In Japan POEM has become the preferred modality for therapy of achalasia due to the excellent results and exceptional safety record. In the US, dedicated POEM devices were approved by the FDA just recently. As a result the bulk of the published data comes from Japan and very little is known regarding outcomes in US population. Therefore the investigators want to prospectively record our experience with POEM as done as part of routine medical care in US population. This will be a data recording study. All patients will receive standard medical care and no experimental interventions will be performed.

DETAILED DESCRIPTION:
Information about the subject's medical history, leading up to the need for an Achalasia treatment, the procedure itself and how the subject does after the procedure, including after the subject gets home, will be collected. This will be done by gathering relevant information from the subject's medical chart and/or by talking with the subject prior to and after the subject's medical procedures. There are no specific study procedures or tests. All information collected is part of the subject's medical care and will be collected even if the subject is not in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Scheduled to undergo POEM treatment

Exclusion Criteria:

* Any contraindication to performing endoscopy
* Participation in another research protocol that could interfere or influence the outcomes measures of the present study.
* The subject is unable/unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those subjects with Achalasia who have been referred for the POEM treatment for their Achalasia.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2013-03; Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Response to POEM treatment | approximately one week
  Information about the subject's medical history, leading up to the need for an Achalasia treatment, the procedure itself and how the subject does after the procedure, including after the subject gets home, will be collected.
  This information will be collected by gathering relevant information from the subject's medical chart and/or by talking with the subject prior to and after the subject's medical procedures.
  There are no specific study procedures or tests. All information collected is part of the subject's medical care and will be collected even if the subject is not in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health, Gainesville, Florida, United States

REFERENCES:
- [Derived] Perbtani YB, Mramba LK, Yang D, Suarez J, Draganov PV. Life after per-oral endoscopic myotomy: long-term outcomes of quality of life and their association with Eckardt scores. Gastrointest Endosc. 2018 Jun;87(6):1415-1420.e1. doi: 10.1016/j.gie.2018.01.019. Epub 2018 Feb 2. PMID 29410304
- [Derived] Pannu D, Yang D, Abbitt PL, Draganov PV. Prospective evaluation of CT esophagram findings after peroral endoscopic myotomy. Gastrointest Endosc. 2016 Sep;84(3):408-15. doi: 10.1016/j.gie.2016.02.022. Epub 2016 Feb 22. PMID 26907745